CLINICAL TRIAL: NCT03045471
Title: The Efficacy and Safety of R-EPOCH and R-CHOP Regimen for Patients With AIDS Associated CD20+ Diffuse Large B Lymphoma
Status: Unknown | Type: Observational
Last Known Status: Not yet recruiting
Sponsor: Shanghai Public Health Clinical Center (Other Government)
Responsible Party: Principal Investigator, Hongzhou Lu, Professor, Shanghai Public Health Clinical Center
Other Study IDs: ARL-1
Record Dates: First submitted 2017-02-03; First posted 2017-02-07 (Estimated); Last update posted 2017-02-07 (Estimated); Status verified 2017-02

CONDITIONS: To Evaluate the Efficacy and Safety of R-EPOCH and R-CHOP Regimen for Patients With AIDS Associated CD20+ Diffuse Large B Lymphoma
MeSH Terms: interventions — Rituximab; R-CHOP protocol

STUDY DESIGN:
Observational Model: Cohort | Time Perspective: Prospective
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: Yes | FDA-regulated Device: No | US Export: No

GROUPS / COHORTS (2):
- R-EPOCH
  Interventions: Drug: R-EPOCH
- R-CHOP
  Interventions: Drug: R-CHOP

INTERVENTIONS:
Drug: R-EPOCH — Rituximab: an anti-CD20 monoclonal antibody, which has the ability to kill B cells, be they normal or malignant; Etoposide: a topoisomerase inhibitor from the group of epipodofyllotoxins; Prednisolone: a glucocorticoid hormone that can cause apoptosis and lysis of both normal and malignant lymphocytes; Oncovin, also known as vincristine: a vinca alkaloid that binds to the protein tubulin, thereby preventing the formation of microtubules and mitosis; Cyclophosphamide: an alkylating antineoplastic agent; Hydroxydaunorubicin, also known as doxorubicin: an anthracycline antibiotic that is able to intercalate DNA, damaging it and preventing the cell division.
  Other Names: Rituximab,Etoposide,Prednisolone,Oncovin,Cyclophosphamide,Hydroxydaunorubici
  Groups: R-EPOCH
Drug: R-CHOP — Rituximab: an anti-CD20 monoclonal antibody, which has the ability to kill B cells, be they normal or malignant; Prednisolone: a glucocorticoid hormone that can cause apoptosis and lysis of both normal and malignant lymphocytes; Oncovin, also known as vincristine: a vinca alkaloid that binds to the protein tubulin, thereby preventing the formation of microtubules and mitosis; Cyclophosphamide: an alkylating antineoplastic agent; Hydroxydaunorubicin, also known as doxorubicin: an anthracycline antibiotic that is able to intercalate DNA, damaging it and preventing the cell division.
  Other Names: Rituximab,Prednisolone,Oncovin,Cyclophosphamide,Hydroxydaunorubici
  Groups: R-CHOP

SUMMARY:
1. Compare the efficacy of R-EPOCH and R-CHOP regimen for patients with AIDS associated CD20+ diffuse large B lymphoma; 2. Compare the safety of R-EPOCH and R-CHOP regimen for patients with AIDS associated CD20+ diffuse large B lymphoma.

ELIGIBILITY:
Inclusion Criteria:

1. male or female aged 18-60 years old;
2. Confirmed as AIDS patients and treated with HAART;
3. Confirmed as CD20+ diffuse large B lymphoma;
4. Serum test; negative for HBV, HCV and syphilis;
5. Hematology: Absolute neutrophil count greater than or equal to 1000/mm(3); Platelet count greater than or equal to 50,000/mm(3); Hemoglobin greater than 8.0 g/dl; Lymphocyte count less than or equal to 4,000/mm(3);
6. Chemistry: Serum ALT/AST less or equal to 5 times the upper limit of normal. Serum creatinine less than or equal to 1.6 mg/dl. Total bilirubin less than or equal to 1.5 mg/dl;
7. Normal cardiac ejection fraction and no evidence of pericardial effusion as determined by an echocardiogram;
8. Negative pregnancy test for female;
9. Patients of both genders must be willing to practice birth control from the time of enrollment on this study and for four months after treatment;
10. To be able to understand and sign the Informed Consent Document with legal force.

Exclusion Criteria:

1. With acute disease, active infection, hemolytic anemia, coagulation dysfunction or diseases of the respiratory, circulation or central nervous system;
2. Patients with heart metastases, CNS metastases or cerebrospinal fluid malignant cells;
3. Women with pregnant or breastfeeding;
4. Any form of primary immunodeficiency;
5. Concurrent Systemic steroid therapy;
6. History of severe immediate hypersensitivity reaction to any of the agents used in this study;
7. History of allogeneic stem cell transplantation.

Ages: 18 Years to 60 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult
Study Population: Patients with AIDS associated CD20+ diffuse large B lymphoma
Sampling Method: Non-Probability Sample
Enrollment: 50 (Estimated)
Dates: Start 2017-03-01 (Estimated); Primary Completion 2020-12-31 (Estimated); Study Completion 2021-12-31 (Estimated)

PRIMARY OUTCOMES:
progression-free survival | 3 years

SECONDARY OUTCOMES:
complete response rate | 3 years
partial response partial response rate | 3 years
overall response | 3 years

IPD SHARING:
Plan to Share IPD: Undecided